CLINICAL TRIAL: NCT00559598
Title: Use of Serum Proteome on the Early Diagnosis of Malignant Biliary-Pancreatic Disease
Brief Title: Blood Proteins in Finding Pancreatic Cancer and Extrahepatic Biliary Tract Cancer
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: 999904272; 04-C-N272; CDR0000573190; NCT00342979 (obsolete NCT alias)
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Extrahepatic Bile Duct Cancer; Pancreatic Cancer
Keywords: pancreatic cancer; extrahepatic bile duct cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Pancreatic Neoplasms

INTERVENTIONS:
Genetic: proteomic profiling
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients with cancer and from healthy participants may help doctors identify and learn more about proteins related to cancer. It may also help doctors tell whether a patient has cancer.

PURPOSE: This clinical trial is looking at proteins in blood samples to see how well they work in finding pancreatic cancer and extrahepatic biliary tract cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To explore the utility of the serum proteome pattern for early detection and diagnosis of pancreatic and extraheptic biliary tract cancer by analyzing serum samples from participants previously enrolled in the PANKRAS-II study.
* To support efforts to contact participants (recruited to the PANKRAS-II study 10 years ago) who were diagnosed with benign biliary-pancreatic disease in order to discern if they subsequently developed a malignant biliary-pancreatic tumor.
* To gather information about clinical factors surrounding the date of blood extraction that may influence the proteomic patterns of the blood samples by performing a review of clinical records of participants.

OUTLINE: Serum samples are analyzed for proteome pattern. Participants undergo a telephone interview about their medical history (i.e., pancreatic or biliary tract disease diagnosed within the past 10 years). Medical records are reviewed to gather information about clinical factors surrounding the date of blood extraction that may influence the proteomic patterns of the blood samples.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Serum samples available from participants meeting any of the following criteria:

  * Diagnosis of pancreatic or extrahepatic biliary tract cancer
  * Suspected of having pancreatic or extraheptic biliary tract cancer, including pathologies (e.g., chronic pancreatitis) that might represent pre-neoplastic stages of the malignant disease
  * Healthy control
* Previously enrolled on the PANKRAS-II study

  * Recruited to study 10 years ago

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2004-08; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Utility of the serum proteome pattern for early detection and diagnosis of pancreatic cancer and extrahepatic biliary tract cancer
Contact participants (recruited to the PANKRAS-II study 10 years ago) who were diagnosed with benign biliary-pancreatic disease in order to discern if they subsequently developed a malignant biliary-pancreatic tumor
Gather information about clinical factors surrounding the date of blood extraction that may influence the proteomic patterns of the blood samples by reviewing clinical records of participants

CONTACTS AND LOCATIONS:
Overall Officials: Lee E. Moore, Principal Investigator — NCI - Occupational and Environmental Epidemiology Branch